CLINICAL TRIAL: NCT00816426
Title: Pharmacokinetics of Standard First and Second Line Anti-TB Drugs in the Lung and Lesions of Subjects Elected for Resection Surgery
Brief Title: Measurement of Anti-TB Drugs in Lung Tissue From Patients Having Surgery to Treat Tuberculosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Korean Center for Disease Control and Prevention (Other Government); International Tuberculosis Research Center (Other); Novartis Institute for Tropical Medicine (Unknown); Asian Medical Center (Unknown)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 999909061; 09-I-N061
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2017-12-29

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Lesions; Pharmacokinetics; Maldistribution; Histopathology
MeSH Terms: conditions — Tuberculosis | interventions — Rifampin; Isoniazid; Pyrazinamide; Kanamycin; Moxifloxacin

ARMS (5):
- 1 (Other): Dosing 2 hours before surgery. -Rifampicin (RIF) will be dosed orally at 600mg or 50mg for subjects under 50kg of bodyweight;-Isoniazid (INH) will be dosed orally at 300mg;-Pyrazinamide (PZA) will be dosed orally at 1.5g;-Moxifloxacin (MXF) will be dosed orally at 400mg;-Kanamycin (KM) will be dosed intramuscularly at 1g or 750mg for subjects under 50kg of body weight
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Kanamycin; Drug: Moxifloxacin
- 2 (Other): Dosing 4 hours before surgery. -Rifampicin (RIF) will be dosed orally at 600mg or 50mg for subjects under 50kg of bodyweight;-Isoniazid (INH) will be dosed orally at 300mg;-Pyrazinamide (PZA) will be dosed orally at 1.5g;-Moxifloxacin (MXF) will be dosed orally at 400mg;-Kanamycin (KM) will be dosed intramuscularly at 1g or 750mg for subjects under 50kg of body weight
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Kanamycin; Drug: Moxifloxacin
- 3 (Other): Dosing 8 hours before surgery. -Rifampicin (RIF) will be dosed orally at 600mg or 50mg for subjects under 50kg of bodyweight;-Isoniazid (INH) will be dosed orally at 300mg;-Pyrazinamide (PZA) will be dosed orally at 1.5g;-Moxifloxacin (MXF) will be dosed orally at 400mg;-Kanamycin (KM) will be dosed intramuscularly at 1g or 750mg for subjects under 50kg of body weight
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Kanamycin; Drug: Moxifloxacin
- 4 (Other): Dosing 12 hours before surgery. -Rifampicin (RIF) will be dosed orally at 600mg or 50mg for subjects under 50kg of bodyweight;-Isoniazid (INH) will be dosed orally at 300mg;-Pyrazinamide (PZA) will be dosed orally at 1.5g;-Moxifloxacin (MXF) will be dosed orally at 400mg;-Kanamycin (KM) will be dosed intramuscularly at 1g or 750mg for subjects under 50kg of body weight
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Kanamycin; Drug: Moxifloxacin
- 5 (Other): Dosing 24 hours before surgery. -Rifampicin (RIF) will be dosed orally at 600mg or 50mg for subjects under 50kg of bodyweight;-Isoniazid (INH) will be dosed orally at 300mg;-Pyrazinamide (PZA) will be dosed orally at 1.5g;-Moxifloxacin (MXF) will be dosed orally at 400mg;-Kanamycin (KM) will be dosed intramuscularly at 1g or 750mg for subjects under 50kg of body weight
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Kanamycin; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Rifampicin — Rifampicin or rifampin (RIF) is a semi-synthetic compound derived from Amycolatopsis rifamycinica. It is mostly used in combination to treat TB, while other disease indications include brucellosis, leprosy, legionnaire's disease and problematic drug-resistant staphylococcal infections. RIF inhibits DNA-dependent RNA polymerase in bacterial cells by binding its beta-subunit, thus preventing transcription to RNA. Its MIC against replicating TB bacilli is 0.1 g/ml and its minimum bactericidal activity (MBC) is 0.5 g/mL. It is one of the rare anti-TB drugs with some activity against nonreplicating cells.
Drug: Isoniazid — Isoniazid (INH) is a first-line antituberculous medication discovered in 1952 and used in the prevention (alone) and treatment (in combination) of tuberculosis. Isoniazid is a prodrug and must be activated by a bacterial catalase to inhibit the synthesis of mycolic acids in the mycobacterial cell wall. Consequently, INH is bactericidal to rapidly-dividing mycobacteria, with an MIC of 0.05 g/ml and an MBC of 1 g/ml, but is inactive if the mycobacterium is nonreplicating or slow-growing.
Drug: Pyrazinamide — Pyrazinamide (PZA) is a synthetic derivative of nicotinamide requiring ctivation by the mycobacterial enzyme pyrazinamidase, only active under acidic conditions which are thought to be found within the phagolysosomal compartment of macrophages. The conversion product, pyrazinoic acid, inhibits fatty acid synthetase I, required by the bacterium to synthesize fatty acids, though this has been disputed. It has an MIC of 6 g/ml and is not cidal under in vitro conditions. Overall, its mechanism of action and reasons for good sterilizing activity in vivo are poorly understood. It is part of the 4-drug combination recommended by the WHO to treat drugsensitive tuberculosis and is also included in most econd-line regimens.
Drug: Kanamycin — Kanamycin (KM) is an aminoglycoside antibiotic belonging to the same class of drugs as Streptomycin, one of the first drugs used to treat TB in the 50 s. It kills sensitive bacteria by binding to the 30S ribosomal subunit and interfering with protein synthesis. Its MIC and MBC against MTB are 2 and 6 g/mL, respectively, with a remarkably low MBC/MIC ratio. However, KM is only used to treat serious bacterial infections due to severe renal toxicity and ototoxicity. No interaction with the metabolism of other drugs has been reported. The drug is approved by the Korean Ministry of Food and Drug Safety (MFDS) but not the US FDA for use against pulmonary TB.
Drug: Moxifloxacin — Moxifloxacin (MXF) is a synthetic fluoroquinolone antibiotic. It inhibits bacterial topoisomerase II (DNA gyrase) and topoisomerase IV, which are essential enzymes playing a crucial role in the replication and repair of bacterial DNA. Its MIC, MBC and intracellular activity against MTB are 0.5, 2 and 1 g/mL, respectively, with again a low MBC/MIC ratio.

SUMMARY:
This study, conducted jointly by researchers at the National Masan TB Hospital, Asan and Samsung Medical Centers in Seoul, Republic of Korea, and the Yonsei University and the NIH in the United States, will examine why some patients with tuberculosis (TB) develop disease that is harder to treat than most cases. TB is an infection of the lung that usually can be successfully treated with anti-TB drugs. However, some people get a more serious kind of disease (called multi-drug resistant TB or extensively drug-resistant TB) that is very difficult to treat and may not be cured by the regular medicines available. This study will try to find out if some of the common TB drugs are getting to the place where the TB bacteria are. It will also look at how current anti-TB drugs might be used more effectively and how better drugs might be developed.

People 20 years of age and older with hard-to-treat TB who have elected to undergo surgical removal of part of their lung at the National Masan Tuberculosis Hospital, Masan, the Asan Medical Center, and the Samsung Medical Center, may be eligible for this study.

Participants undergo the following procedures:

* Medical history and physical examination, including sputum sample.
* Blood tests at various times during the study.
* Drug administration. Subjects are given one dose each of five common TB drugs rifampicin, isoniazid, pyrazinamide, kanamycin and moxifloxacin before they undergo surgery to remove part of their lung. After surgery, some of the lung tissue and fluid around the lungs that was removed during surgery will be examined to determine the regions where the TB bacteria live and analyze the lung tissue itself.
* Dynamic MRI (magnetic resonance imaging) scan. This type of scan uses a magnetic field and radio waves to produce pictures of the lung. Subjects lie very still on a table inside the cylindrical scanner with their head on a soft cradle and their hands over their head. Several images are obtained for less than 5 minutes at a time.

DETAILED DESCRIPTION:
It takes 6 to 24 months of intensive combination therapy to cure tuberculosis (TB) with antibiotics that have proven activity in vitro. In contrast, many pulmonary infectious diseases can be cured following single drug treatment with similar drugs for only one to a few weeks. We hypothesize that the unusual complexity of TB lesions and the degree of sequestration of TB bacilli within these lesions may limit access of the drugs to their site of action, leading to treatment failure, long treatment duration and the emergence of drug resistance. To test the hypothesis that drug maldistribution into lesions impacts on treatment duration and failure, we propose to examine the lesion-specific penetration properties of 5 standard anti-TB drugs in the lungs of subjects selected for lung surgery. The study is designed to understand what lesion types are the most difficult to penetrate. This aspect of TB drug pharmacokinetics has been largely neglected so far, probably owing to the lack of adequate technology and the limited availability of human TB lesion samples. Fifteen patients who elect lung resection surgery will be asked to participate in the study. Consented subjects will receive 4-5 first and second line anti-TB drugs concomitantly at 1 of 5 pre-determined times prior to surgery. At the time of resection, drug levels will be measured in plasma, in uninvolved lung tissue and in lesions using standard analytical methods as well as imaging Mass Spectrometry (MS) where drug concentration gradients can be visualized across tissue sections. The major aim of this study is to determine actual concentrations and permeability coefficients of the 5 study drugs in various lesion types contained within subjects surgically removed lung tissue. Data analysis will also provide the relative exposure of each drug in plasma versus lung tissue and lesion. If conclusive, the results may be taken into consideration when selecting drug doses and dosing regimens. Additionally, images generated by standard of care (SOC) High Resolution Computed Tomography (HRCT), and Dynamic MRI for each subject will provide information regarding lesion structure and anatomy, lesional blood flow and microvascular function. Lesion-specific correlations will be established between CT radiology and drug pharmacokinetic (PK) to identify which histopathologic lesion types may be particularly difficult to sterilize and to evaluate the potential impact of drug penetration on treatment outcome. The long term goal of this study is to identify the factors behind poor lesion penetration, so that new agents can be optimized with better penetration properties to target harder-to-sterilize lesion' types.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Males and females age 20 and above
  2. Selected for lung resection due to anti-tuberculous treatment failure, multidrug resistant disease, or other reason determined by the treating physician
  3. Radiographic evidence of tuberculous disease of the lung(s)
  4. If already on an aminoglycoside, ability and willingness to substitute this aminoglycoside with KM for the one study dose
  5. Willingness to receive MRI scan and marker and Gadolinium injection
  6. Willingness to have samples stored
  7. Ability and willingness to give written or oral informed consent

EXCLUSION CRITERIA:

1. Subjects less than 20 years of age
2. Women of childbearing potential who are pregnant, breast feeding, or unwilling to avoid pregnancy (i.e., the use of appropriate contraception including oral and subcutaneous implantable hormonal contraceptives, condoms, diaphragm, intrauterine device (IUD), or abstinence from sexual intercourse) [Note: Prospective female participants of childbearing potential must have negative pregnancy test (urine) within 48 hours prior to study entry.]
3. Allergy or hypersensitivity to any of the 5 study drugs, any aminoglycoside, or rifamycin (those allergic to fluoroquinolones will not receive MXF).
4. Those with severe gout
5. Severe claustrophobia or Gadolinium hypersensitivity (tbc)
6. Renal, hepatic, auditory and/or vestibular impairment.

   1. Serum creatinine greater than 2.0 mg/dL (renal)
   2. Aspartate aminotransferase (AST or SGOT) greater than 100 IU/L (LFTs)
   3. Alanine aminotransferase (ALT or SGPT) greater than 100 IU/L (LFTs)
   4. Total bilirubin greater than 2.0 mg/dL (LFTs)
7. The use of any of Rifampicin (RIF), Rifapentine or Rifabutin within 30 days prior to the study
8. HIV infection, determined by a positive HIV test performed with the past 6 months
9. The use of any of the following drugs within 30 days prior to study:

   1. Systemic cancer chemotherapy
   2. Systemic corticosteroids (oral or IV only) with the following

      exceptions (i.e.the following are NOT exclusion criteria): intranasal, topical, and inhaled corticosteroids, a short course (10 days or less) of corticosteroids for a non-chronic condition completed at least 2 weeks prior to enrollment in this study
   3. Systemic IND agents other than Linezolid
   4. Antiretroviral medications
   5. Growth factors
10. The need for ongoing therapy with warfarin, phenytoin, lithium cholestrymine, levodopa, cimetidine, disulfiram, ergot derivatives, fosphenytoin, carbamazepine, cyclosporine, tacrolimus, sirolimus, amiodarone or Phenobarbital (If a potential subject is on one of these medications but it is being stopped per standard of care, to be eligible for the study the drug must be stopped at least one day prior to receiving study drug. A longer washout period is not necessary.) The only exception to this is amiodarone; because of amiodarone s long half-life and potential for QT prolongation, it should be stopped at least 60 days prior to receiving study drugs.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12-29; Primary Completion 2014-08-26 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Comparison between the relative permeability coefficients of RIF and KM in pathologically defined large caseous necrotic nodules. | Dosing given 24 hours- 2 hours before surgery

SECONDARY OUTCOMES:
The comparison between the relative permeability coefficients of RIF, KM, INH, PZA and MXF in caseous necrotic nodules versus open cavities | Dosing given 24 hours -2 hours before surgery, then endpoint assessed from time of surgery.
The comparison between the absolute permeability coefficients of each of the five drugs in uninvolved lung and in closed necrotic lesions | Dosing given 24 hours -2 hours before surgery, then endpoint assessed from time of surgery.
The comparison between the exposure ratio or ratio between the Area Under the Curve (AUC0-24) in lesions (AUClesion), uninvolved lung (AUClung) and plasma (AUCplasma) for RIF and KM in large caseous necrotic nodules | Dosing given 24 hours -2 hours before surgery, then endpoint assessed from time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- South Korea (3):
  - Pusan National Unversity Hospital (PNUH), Busan
  - Asan Medical Center, Seoul
  - National Medical Center, Seoul

REFERENCES:
- [Background] Soman A, Honeybourne D, Andrews J, Jevons G, Wise R. Concentrations of moxifloxacin in serum and pulmonary compartments following a single 400 mg oral dose in patients undergoing fibre-optic bronchoscopy. J Antimicrob Chemother. 1999 Dec;44(6):835-8. doi: 10.1093/jac/44.6.835. PMID 10590288
- [Background] Drexler DM, Garrett TJ, Cantone JL, Diters RW, Mitroka JG, Prieto Conaway MC, Adams SP, Yost RA, Sanders M. Utility of imaging mass spectrometry (IMS) by matrix-assisted laser desorption ionization (MALDI) on an ion trap mass spectrometer in the analysis of drugs and metabolites in biological tissues. J Pharmacol Toxicol Methods. 2007 May-Jun;55(3):279-88. doi: 10.1016/j.vascn.2006.11.004. Epub 2006 Dec 5. PMID 17222568
- [Background] Wagner C, Sauermann R, Joukhadar C. Principles of antibiotic penetration into abscess fluid. Pharmacology. 2006;78(1):1-10. doi: 10.1159/000094668. Epub 2006 Jul 19. PMID 16864973
- [Derived] Strydom N, Gupta SV, Fox WS, Via LE, Bang H, Lee M, Eum S, Shim T, Barry CE 3rd, Zimmerman M, Dartois V, Savic RM. Tuberculosis drugs' distribution and emergence of resistance in patient's lung lesions: A mechanistic model and tool for regimen and dose optimization. PLoS Med. 2019 Apr 2;16(4):e1002773. doi: 10.1371/journal.pmed.1002773. eCollection 2019 Apr. PMID 30939136